CLINICAL TRIAL: NCT02838784
Title: The Efficacy and Safety of Artacent™ for Treatment Resistant Lower Extremity Venous and Diabetic Ulcers: A Prospective Randomized Study
Brief Title: Efficacy and Safety of Artacent™ for Treatment Resistant Lower Extremity Venous and Diabetic Ulcers
Acronym: TMArtacent
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tides Medical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 16-001
Record Dates: First submitted 2016-07-15; First posted 2016-07-20 (Estimated); Last update posted 2017-10-13 (Actual); Status verified 2017-10

CONDITIONS: Venous Ulcer; Foot Ulcer, Diabetic
MeSH Terms: conditions — Varicose Ulcer; Diabetic Foot | interventions — Standard of Care; Debridement

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Artacent Human Amniotic Membrane (Experimental): Patients randomized to the Artacent group will receive standard of care (off-loading with a removable cast walker and non-adherent dressings in addition to debridement and use of moisture retentive dressing) and the application of the Artacent amniotic allograft once every two weeks for up to 5 applications or until the ulcer has healed.
  Interventions: Other: Artacent Human Amniotic Membrane
- Lower Extremity Ulcer Standard of Care (Active Comparator): Patients randomized to standard of care will receive off-loading with a removable cast walker and non-adherent dressings (e.g. Adaptic) in addition to debridement and use of moisture retentive dressings. An outer dressing will also be applied.
  Interventions: Procedure: Standard of Care

INTERVENTIONS:
Other: Artacent Human Amniotic Membrane — Double layer dehydrated amnion product
  Other Names: Amniotic tissue allograft; Amniotic placental membranes
  Arms: Artacent Human Amniotic Membrane
Procedure: Standard of Care — Off loading with a cast walker, non-adherent dressings, debridement and moisture retentive dressings
  Other Names: Debridement; Off-loading; non-adherent dressings
  Arms: Lower Extremity Ulcer Standard of Care

SUMMARY:
This study will compare the proportion of patients who have wound closure within 12 weeks as well as the time to wound closure in patients receiving Artacent™ versus standard of care for treatment of non-healing lower extremity wounds. The recurrence of healed wounds will be assessed at 6 months via a telephone survey

DETAILED DESCRIPTION:
This study is to document the efficacy of Artacent™ Human Amniotic Membrane (Artacent) in the treatment of diabetic and vascular lower extremity ulcers. The study will add to the currently available literature by also assessing the impact of treatment on quality of life and on heal economic outcomes. Finally the study will follow patients for longer than previous studies and will obtain data on healing and recurrence at 6 months.

The objectives of this study are 1) to compare Artacent to standard of care (SOC) in the treatment of non-healing lower extremity ulcers and 2) to evaluate the impact of treatment on patient quality of life. Health economic outcomes will also be collected. The proportion of patients receiving Artacent who have wound closure with 12 weeks will be compared to those patients receiving SOC only will be compared. A comparison of time to wound closure will also be compared between the two populations.

Patients who are randomized to the SOC group (control) and require further treatment at 12 weeks due to incomplete wound healing, may receive treatment with Artacent if the investigator determines that to be a potentially beneficial option.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Able and willing to give consent and to comply with study
* Lower extremity ulcer between 1 and 25 cm2 point after the 4 week run-in period
* Has received documented SOC treatment for 4 weeks or greater duration resulting in <50% reduction in the ulcer size
* No clinical signs of infection at the ulcer site
* Serum Creatinine below 3.0 mg/dl
* Serum HgA1c below 12%
* Adequate circulation to the affected limb with ABI between 0.7 and 1.2 or tri-/bi-phasic arterial waveforms at the ankle of the affected leg.

Exclusion Criteria:

* Is participating in another wound study
* Has a Charcot foot
* Has previously received a different biological graft on the target foot
* Has more than one lower extremity ulcer
* Has an ulcer that probes to bone or involves tendon, muscle, joint capsule or has sinus tracts
* Is currently receiving radiation or chemotherapy
* Has an autoimmune connective tissue disorder
* Is taking any medication known to be an immune system modulator
* Is pregnant or is considering becoming pregnant within the next 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2016-09; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Wound closure | 12 weeks
  100% re-epithelialization of the wound without drainage or need for use of a dressing
Time to wound closure | 12 weeks
  # of days to 50% or greater closure
Ulcer recurrence | 6 months
  Telephone survey to capture number of ulcer recurrences and treatment

SECONDARY OUTCOMES:
Quality of Life | 12 weeks
  EQ-5D survey
Impact of Treatment on Return to Work | 12 weeks
  Employment status e.g. full-time, part-time, retired, unemployed, etc.
Time to full weight bearing status | 12 weeks
  Ability of the subject to bear full weight and the time to full weight bearing
Adverse Events and Secondary Treatments | 12 weeks
Number of grafts and graft size(s) | 12 weeks
  Number and size of grafts used at each application will be collected.

OTHER OUTCOMES:
Health economic outcomes | 12 weeks
  Collection of de-identified Explanation of Benefits (EOB) and/or submitted claims and/or documentation of procedures via CPT coding.

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Global Podiatry Partners, Inc, Arcadia, California
  - Iberia Medical Center, New Iberia, Louisiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Foot & Ankle Center of Nebraska, Omaha, Nebraska
  - Livingston Podiatry Associates PLLC, Bellmore, New York
  - Foot & Ankle Physicians of Ohio, Grove City, Ohio
  - Southwest Austin Foot & Ankle Clinic, PLLC, Austin, Texas

IPD SHARING:
Plan to Share IPD: Undecided